CLINICAL TRIAL: NCT02763995
Title: Pharmacotherapy Follow-up in Older HIV-infected Patients: Impact on Cardiovascular Risk and Quality of Life
Brief Title: Pharmacotherapy Follow-up in Older HIV-infected Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elza Aparecida Machado Domingues (Other)
Responsible Party: Sponsor-Investigator, Elza Aparecida Machado Domingues, MSc, Universidad de Granada
Organization: Universidad de Granada (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: University of Granada
Record Dates: First submitted 2016-04-27; First posted 2016-05-05 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: HIV
Keywords: HIV; pharmaceutical care; older patients; cardiovascular risk; pharmacotherapy follow up
MeSH Terms: interventions — Pharmaceutical Services

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pharmaceutical care (Experimental): Dader method. Health education for lifestyle modification. Improve adherence. Resolution of negative outcome associated with medication.
  Interventions: Behavioral: Pharmaceutical care

INTERVENTIONS:
Behavioral: Pharmaceutical care — This is a quasi-experimental study and the same group will be evaluated before and after the follow up.

SUMMARY:
Cardiovascular diseases (CVD) are the main cause of death in Spain. In HIV patients, the uncontrolled viral replication, antiretroviral therapy (ART) and coinfections contribute to develop metabolic diseases and increase the prevalence of risk factors for CVD. These patients are aging which results in a higher probability of comorbidities, increased number of medications, possibility of having a negative outcome associated with medication (NOM) and increased cardiovascular risk (CVR). Various studies have established that pharmaceutical care (PC) results in better control of cardiovascular risk factors.

The purpose of this study is to evaluate the impact of pharmaceutical care achieved through pharmacotherapy follow-up on cardiovascular risk and health related quality of life (HRQoL) of HIV patients older than 50.

DETAILED DESCRIPTION:
Quasi-experimental clinical study, pre-post intervention, performed with one patient cohort.

Study will be carry out at a tertiary hospital. The population will be constituted of patients who receive care from the outpatient department of the pharmacy service in use of antiretroviral therapy.

Variables will be obtained from patients' clinical histories, from dispensing records and through interviews with patients.

Main variables:

* cardiovascular risk estimated according to Systematic Coronary Risk Evaluation (SCORE) and Registre Gironí del Cor (REGICOR) equations
* HRQoL measured by the Short-Form 36-Item Health Survey (SF-36) and Medical Outcomes Study HIV Health Survey (MOS-HIV) questionnaires.

Other variables: sociodemographic, clinical, pharmacological, related to CVR, related to NOM and to the interventions.

Interventions will be performed every two months until complete 12 months of follow-up. Pharmacotherapy follow-up will be conducted according to the Dader method. The interventions will be health education for lifestyle modification, improve adherence and aimed to the resolution of NOM and drug-related problems.

ELIGIBILITY:
Inclusion Criteria:

* patients older than 50 years
* in use of antiretroviral therapy
* cardiovascular risk ≥2%, estimated by the SCORE equation
* accept to participate in the research through the signature of a written informed consent

Exclusion Criteria:

* patients with neurodegenerative deficit or HIV dementia
* participants in clinical trials
* non signature of a written informed consent

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-04; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Cardiovascular risk estimation | Baseline and 12 months
  Change in cardiovascular risk estimated by SCORE equation will be evaluated after one year of Pharmaceutical Care
Cardiovascular risk estimation | Baseline and 12 months
  Change in cardiovascular risk estimated by REGICOR equation will be evaluated after one year of Pharmaceutical Care
Health-related quality of life | Baseline and 12 months
  Change in health-related quality of life measured by SF-36 questionnaire will be evaluated after one year of Pharmaceutical Care.
Health-related quality of life | Baseline and 12 months
  Change in health-related quality of life measured by MOS-HIV questionnaire will be evaluated after one year of Pharmaceutical Care.

SECONDARY OUTCOMES:
Systolic and diastolic blood pressure | Baseline and 12 months
  Change in systolic and diastolic blood pressure will be evaluated after one year of Pharmaceutical Care
Total cholesterol levels | Baseline and 12 months
  Change in total cholesterol levels will be evaluated after one year of Pharmaceutical Care
High-density lipoprotein (HDL-c) levels | Baseline and 12 months
  Change in HDL-c will be evaluated after one year of Pharmaceutical Care
Low-density lipoprotein (LDL-c) levels | Baseline and 12 months
  Change in LDL-c will be evaluated after one year of Pharmaceutical Care
Triglycerides levels | Baseline and 12 months
  Change in triglycerides levels will be evaluated after one year of Pharmaceutical Care
Glucose levels | Baseline and 12 months
  Change in glucose levels will be evaluated after one year of Pharmaceutical Care
Number of patients with smoking cessation | Baseline and 12 months
  Patients that achieve smoking cessation after one year of Pharmaceutical Care

CONTACTS AND LOCATIONS:
Overall Officials: Elza Aparecida M Domingues, MSc, Principal Investigator — Universidad de Granada; Miguel Angel Calleja Hernandez, PhD, Study Director — University Hospital Virgen de las Nieves; Monica Ferrit Martin, PhD, Study Director — University Hospital Virgen de las Nieves
Locations (1):
- Hospital Universitario Virgen de las Nieves, Granada, Spain

IPD SHARING:
Plan to Share IPD: Undecided